CLINICAL TRIAL: NCT07361588
Title: Feasibility Study for VCool™ Intranasal Cooling System in Healthy Volunteers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NeuroIntact Inc. (Industry)
Collaborators: University of Maryland, Baltimore (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Bryan Wand, Director of Engineering, NeuroIntact Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 00080424; M6785424C6544 (Other Grant/Funding Number: MARCORSYSCOM- Marine Corps System Command - Department of defense)
Record Dates: First submitted 2025-12-31; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Targeted Temperature Management
Keywords: targeted temperature management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Healthy adult volunteers (Experimental): The study is designed to gather preliminary data regarding air flow rates and time required to reduce core body temperature to 35.5℃ and maintain the temperature between 35℃ and 36℃ for one hour after cooling.
  Interventions: Device: Targeted Temperature Management Intranasal Cooling System

INTERVENTIONS:
Device: Targeted Temperature Management Intranasal Cooling System — VCool Intranasal Cooling System

SUMMARY:
The objective of this study is to evaluate the performance and safety of the VCool Intranasal Cooling System in healthy adult volunteers. The study is designed to gather preliminary data regarding air flow rates and time required to reduce core body temperature to 35.5℃ and maintain the temperature between 35℃ and 36℃ for one hour after cooling.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ages 18 to 55.
2. An Institutional Review Board (IRB) approved informed consent is signed and dated prior to any study-related activities.
3. Baseline core body temperature between 36.8℃ and 37.5℃.
4. Have the ability to understand the requirements of the study and are willing to comply with all study procedures.
5. In the opinion of the Investigator, are able to participate in the study.

Exclusion Criteria:

1. History of cardiovascular, respiratory, or metabolic disorder
2. Any contraindication to undergoing Magnetic Resonance Imaging (MRI)
3. Pregnant
4. Severe peripheral vascular disease
5. History of Raynaud's disease
6. Currently experiencing a respiratory infection
7. Chronic rhinosinusitis
8. History of sickle cell disease
9. History of cold agglutinin disease
10. History of cryoglobulinemia
11. Known deviated septum or nasal deformity
12. History of nosebleeds or a nosebleed within past 24 hours
13. Use of antipyretics or other medications affecting body temperature within the past 24 hours.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
lower core body temperature | 1 hour
  To confirm the VCool System can lower core body temperature to 35.5℃.
maintain a core body temperature | 1 hour
  To confirm the VCool System can maintain a core body temperature between 35℃ and 36℃ for one hour after cooling.
differential between core body and brain temperature | 2 hours
  To evaluate the differential between core body and brain temperature while using VCool.

SECONDARY OUTCOMES:
Bedside Shivering Assessment Scale (BSAS). | 2 hours
  To assess the shivering experienced by participants based on the 4-point Bedside Shivering Assessment Scale (BSAS).

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Badjatia, MD, MS, Study Chair — University of Maryland
Locations (1):
- R Adams Cowley Shock Trauma Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2025-11-25): https://cdn.clinicaltrials.gov/large-docs/88/NCT07361588/Prot_000.pdf
  • Informed Consent Form (2025-12-12): https://cdn.clinicaltrials.gov/large-docs/88/NCT07361588/ICF_001.pdf